CLINICAL TRIAL: NCT01259999
Title: Distribution of an Energy Rich Formula at Medication Rounds to Individuals Living in Old Peoples Home - Effects on Energy Intake Compared to Standard Nutritional Treatment
Brief Title: Energy Dense Formula to People Living in Old Peoples Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Gerd Faxén Irving, Karolinska University Hospital Huddinge and Karolinska Institutet/NVS
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Huddinge Municipality and SLL
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Protein-Energy Malnutrition; Anorexia; Weight Change
Keywords: malnutrition; oleic-acid; micronutrient supplement; old peoples home
MeSH Terms: conditions — Protein-Energy Malnutrition; Anorexia; Body Weight Changes; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Energy dense formula (Experimental)
  Interventions: Dietary Supplement: Calogen extra strawberry

INTERVENTIONS:
Dietary Supplement: Calogen extra strawberry — A daily dose of 3 x 30 ml Calogen extra strawberry flavour will be distributed at the same time as the medicines i.e. at 8.00, 12.00 and 20.00.
  Other Names: Nutricia PDS:1005912

SUMMARY:
Dietary intake in frail elderly is often lower than estimated needs due to the combined effects of the anorexia of ageing, frailty and the presence of acute and chronic disease. The objectives of the present study are to assess the effects of an oleic acid rich formula fortified with micronutrients on energy intake, vitamin- and mineral status, muscle strength and mobility. The investigators have recently performed a similar study in an acute ward setting without micronutrients.

DETAILED DESCRIPTION:
Malnutrition has been reported to be present in up to 55% of acutely hospitalised elderly and in one third of people living in assisted accommodation. Frail elderly with poor appetite are at risk for malnutrition. Rebecca Stratton et al have reviewed effects of oral nutritional supplements (ONS) in elderly hospital patients and key findings in hospital trials were that ONS can improve intakes of energy, protein and micronutrients without substantially reducing food intake which may lead to weight gain or attenuate weight loss.

Calogen extra is a fat emulsion containing 400 kcal/100 ml, based on canola and sunflower-oil which has a good fat composition. Moreover it contains around 30 % of recommended micronutrients and 5g protein/100 ml. It has potentially positive effects on energy intake, fatty acid profile and constipation.

The investigators have recently performed a clinical trial in geriatric patients in an acute-ward setting to evaluate the effects of a similar fat emulsion, Calogen, without micronutrients. The investigators could conclude that this fat emulsion based on MUFA and PUFA distributed three times daily at medication rounds may have positive effects on weight, appetite and serum lipids. Moreover the approach was well accepted by patients and nurses. The intervention period was very short (median 8 days) therefore the investigators plan to perform a study with a similar design, for a longer period of time, in a group of elderly living in old peoples home.

ELIGIBILITY:
Inclusion Criteria:

* >65 years old
* Mini nutritional assessment-short form (MNA-SF)score < 12 points
* able to give informed consent.

Exclusion Criteria:

* pancreatitis
* fat malabsorption, non-consent for participation.
* Subjects that have Calogen will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Increased intake of energy and nutrients | 6 weeks as intervention 6 weeks as control
  The sample size has been estimated upon a minimum difference in daily energy intake between the Control and Calogen group of 200 kcal (4). To detect a significant difference in energy intake at the 5% significance level and with 80% power 27 subjects in each group were needed. To allow for study drop-outs this is increased to 30 subjects in each group.

SECONDARY OUTCOMES:
Increased appetite | 6 weeks intervention 6 weeks control

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Faxen Irving, RD, PHD, Principal Investigator — Karolinska University Hospital Huddinge/NVS/KI
Locations (1):
- Dep of Geriatrics, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Tylner S, Cederholm T, Faxen-Irving G. Effects on Weight, Blood Lipids, Serum Fatty Acid Profile and Coagulation by an Energy-Dense Formula to Older Care Residents: A Randomized Controlled Crossover Trial. J Am Med Dir Assoc. 2016 Mar 1;17(3):275.e5-11. doi: 10.1016/j.jamda.2015.12.005. Epub 2016 Jan 23. PMID 26810442